CLINICAL TRIAL: NCT05747807
Title: Percutaneous Intradiscal Radiofrequency as A Treatment for Radicular Pain From Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Rarinthorn Choomsai Na Ayuthaya, MD, Principal Investigator, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0120/66
Record Dates: First submitted 2023-02-08; First posted 2023-02-28 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Disk Herniated Lumbar; Radicular Pain; Intradiscal Radiofrequency

STUDY DESIGN:
Intervention Model Description: One group pre-posttest design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Percutaneous intradiscal radiofrequency (Experimental): Standard monitoring ,prone position, sterile prepped and draped No sedation, Fentanyl 0.5-2 mcg/kg IV as needed ATB prophylaxis: ceftriaxone 1 g IV Performed by interventional pain physician, under fluoroscopic guidance 2% lidocaine 5 ml LA using Flextrode introducer kit, Boston Scientific Corporation Using an extrapedicular approach ipsilateral to the prolapse, the Flextrode cannula is advanced to the posterior disc.
  The Flextrode electrode is inserted through the cannula. Sensory (50Hz) and motor (2Hz) stimulation, 3 Volts amplitude and 1msec pulse width. Confirm no sensory/motor response.
  Lateral, AP, and oblique x-ray views are used to confirm the active tips are fully within the disc Thermal RF: temp 80 ◦C, 4 min Ceftriaxone 75 mg intradiscal injection via the cannula
  Interventions: Device: Percutaneous intradiscal radiofrequency treatment

INTERVENTIONS:
Device: Percutaneous intradiscal radiofrequency treatment — using heat created by radiofrequency electrode to destroy the nociceptive pain fibres and enhance the structural integrity of the disc
  Other Names: Flextrode

SUMMARY:
The goal of this clinical trial is to demonstrate the efficacy of percutaneous intradiscal radiofrequency as a treatment for radicular pain from lumbar disc herniation.

The main question it aims to answer is:

• Can percutaneous intradiscal radiofrequency lower the severity of radicular pain from lumbar disc herniation Participants will be treated with percutaneous intradiscal radiofrequency and evaluated for radicular pain severity before and 3 months after the procedure.

There is no comparison group.

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 year-old patients with radicular pain from lumbar disc herniation for ≥ 3 months
2. Lumbar disc herniation ≤ 2 locations evidenced by MRI, with ≥ 50% remaining disc height, without disc sequestration
3. Previously treated with epidural steroid injection (ESI) and achieved ≥ 50 % pain relief from local anesthetic effect, confirming radicular pain from lumbar disc herniation, but did not respond to ESI (< 50 % Pain relief or pain relief < 3 months)

Exclusion Criteria:

* Patient refusal
* Discitis
* Previous lumbar spine surgery
* Progressive neurological deficit and/or cauda equina syndrome
* Coagulopathy
* Allergic to any medication in study protocols
* Unable to rate the pain
* Pain in any area worse than the radicular pain

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline radicular pain score at 2 weeks | pre-treatment and 2 week post-treatment
  Radicular pain severity using numerical rating scale (0-10) Zero represents 'no pain at all' whereas 10 represents 'the worst pain ever possible'.
Change from baseline radicular pain score at 3 months | pre-treatment and 3 months post-treatment
  Radicular pain severity using numerical rating scale (0-10) Zero represents 'no pain at all' whereas 10 represents 'the worst pain ever possible'.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) at baseline | pre-treatment
  using Oswestry questionnaire version 1.0 - Thai version
  The ODI is comprised of 10 questions that ask patients about their ability to manage everyday life, and covers intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question contains 6 statements that correlate to a score of 0 through 5, where the patient is to choose the statement that best matches their ability. To obtain the index, the scores of all questions are summed and then multiplied by two.
  The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Oswestry Disability Index (ODI) at 2 weeks | 2 week post-treatment
  using Oswestry questionnaire version 1.0 - Thai version
  The ODI is comprised of 10 questions that ask patients about their ability to manage everyday life, and covers intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question contains 6 statements that correlate to a score of 0 through 5, where the patient is to choose the statement that best matches their ability. To obtain the index, the scores of all questions are summed and then multiplied by two.
  The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
  using Oswestry questionnaire version 1.0 - Thai version
Oswestry Disability Index (ODI) at 3 months | 3 month post-treatment
  using Oswestry questionnaire version 1.0 - Thai version
  The ODI is comprised of 10 questions that ask patients about their ability to manage everyday life, and covers intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question contains 6 statements that correlate to a score of 0 through 5, where the patient is to choose the statement that best matches their ability. To obtain the index, the scores of all questions are summed and then multiplied by two.
  The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
  using Oswestry questionnaire version 1.0 - Thai version
WHOQOL-Brief total score at baseline | pre-treatment
  using WHOQOL-Brief-Thai questionnaire
  The WHO Quality of Life-BREF (WHOQOL-BREF) is a 26-item questionnaire that measures an individual's quality of life.
  The final score ranges from 0-100. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health.
WHOQOL-Brief total score at 2 weeks | 2 week post-treatment
  using WHOQOL-Brief-Thai questionnaire
  The WHO Quality of Life-BREF (WHOQOL-BREF) is a 26-item questionnaire that measures an individual's quality of life.
  The final score ranges from 0-100. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health.
WHOQOL-Brief total score at 3 months | 3 month post-treatment
  using WHOQOL-Brief-Thai questionnaire
  The WHO Quality of Life-BREF (WHOQOL-BREF) is a 26-item questionnaire that measures an individual's quality of life.
  The final score ranges from 0-100. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No